CLINICAL TRIAL: NCT07253324
Title: A Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ENX-104 in Participants With Major Depressive Disorder With Anhedonia
Brief Title: ENX-104 MAD Study for Participants With Major Depressive Disorder With Anhedonia (aMDD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Engrail Therapeutics INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENX-104-003
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENX-104 (Experimental)
  Interventions: Drug: ENX-104
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ENX-104 — Oral Solution
  Arms: ENX-104
Drug: Placebo — Oral solution
  Arms: Placebo

SUMMARY:
The study is designed to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of ENX-104 in participants with major depressive disorder with anhedonia (aMDD).

ELIGIBILITY:
Inclusion Criteria:

* Biologically female participants (defined as assigned female at birth)

  1. Of non-childbearing potential, defined as either permanently sterilized or postmenopausal and with a negative pregnancy test.
  2. Of childbearing potential and willing to use both a highly effective method of contraception and a condom with any partner or remain abstinent, and with a negative pregnancy test
  3. Not currently breastfeeding or lactating, and not intending to initiate breastfeeding during the course of study conduct
* Biologically male participants (defined as assigned male at birth), if fertile must be willing to have a partner use a highly effective method of contraception and participant use a condom with any partner of childbearing potential, or remain abstinent

Exclusion Criteria:

* Unable or unwilling to comply with the requirements of the study or, in the opinion of the Investigator or Sponsor, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-11-26 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAE) | From Day 1 up to Day 21

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - MAC Clinical Research, Blackpool, Lancashire
  - MAC Clinical Research, Prescot, Merseyside
  - MAC Clinical Research, Cannock, South Staffordshire
  - MAC Clinical Research, Manchester

IPD SHARING:
Plan to Share IPD: No